CLINICAL TRIAL: NCT03843541
Title: A Phase III, Multi-centre, Randomized, Rater- and Patient-blind, Placebo- and Active-controlled, Parallel Group Clinical Trial to Compare the Efficacy and Safety of 1-week Treatment of Intravenous N-acetylcysteine (NAC) 600 mg Twice Daily (Active Test Treatment), Ambroxol Hydrochloride 30 mg Twice Daily (Active Control Treatment) and Placebo as Expectorant Therapies in Adult Chinese Patients With Respiratory Tract Diseases and Abnormal Mucus Secretions
Brief Title: A Clinical Trial to Compare the Efficacy and Safety of 1-week Treatment of Intravenous N-acetylcysteine (NAC) 600 mg Twice Daily, Ambroxol Hydrochloride 30 mg Twice Daily and Placebo as Expectorant Therapies in Adult Chinese Patients With Respiratory Tract Diseases and Abnormal Mucus Secretions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z7244L01
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Tract Diseases; Abnormal Mucus Secretions
Keywords: N-acetylcysteine (NAC); ambroxol hydrochloride; bronchitis; cystic fibrosis; fibrosis bronchiectasis; increased sputum viscosity; cough; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Respiratory Tract Diseases; Bronchitis; Cystic Fibrosis; Cough; Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine; Ambroxol

STUDY DESIGN:
Intervention Model Description: There will be 3 treatment groups of NAC, ambroxol and placebo. A total of 333 patients will be randomized to NAC or ambroxol or placebo in a 1:1:1 ratio. Approximately 111 patients will be randomized in each treatment group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both rater and patient will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active test treatment-NAC (Experimental): NAC 600mg will be administered by slow intravenous infusion twice daily for the 1-week treatment period.
  Interventions: Drug: N-acetylcysteine (NAC) 600 mg
- Active control treatment-Ambroxol hydrochloride (Active Comparator): Ambroxol hydrochloride 30 mg will be administered by slow intravenous infusion twice daily for the 1-week treatment period.
  Interventions: Drug: Ambroxol hydrochloride 30 mg
- Placebo (Placebo Comparator): Placebo will be administered by slow intravenous infusion twice daily for the 1-week treatment period.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) 600 mg — NAC will be administered twice a day, morning and evening, during treatment period.
  Other Names: Fluimucil®
  Arms: Active test treatment-NAC
Drug: Ambroxol hydrochloride 30 mg — Ambroxol hydrochloride will be administered twice a day, morning and evening, during treatment period.
  Other Names: Mucosolvan®; Fluibron®
  Arms: Active control treatment-Ambroxol hydrochloride
Other: placebo — Placebo will be administered twice a day, morning and evening, during treatment period.
  Arms: Placebo

SUMMARY:
This is a phase 3, multicenter, randomized, rater- and patient-blind, placebo- and active-controlled, 3-arm parallel group clinical trial. Patients will be randomized to N-acetylcysteine (NAC) or ambroxol or placebo in a 1:1:1 ratio. A total of approximately 333 patients in China will be randomized. The total study duration will be approximately 8 months including the enrolment period of approximately 7 months and the patient participation duration of 1 month or 4 weeks. Each patient will undergo a screening period of up to 1 week, a 1-week treatment period and a 2-week follow-up period. This study will be conducted in approximately 15-25 sites in China.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult (≥18 years old) hospitalized patients with respiratory tract diseases and abnormal mucus secretions such as: acute bronchitis, chronic bronchitis and exacerbations, emphysema, mucoviscidosis and bronchiectasis.
2. Chinese ethnicity and/or Chinese
3. Signed the informed consent form before any study-related procedure
4. Sputum viscosity score ≥ 2 at randomization visit
5. Expectoration difficulty score ≥ 2 at randomization visit
6. Willingness and ability to comply with study procedures

Exclusion Criteria:

1. Intolerance or contra-indication to treatment with NAC or ambroxol or allergy to any component of the study treatments
2. (For female patients) ongoing pregnancy or lactation, or childbearing potential but unwillingness to adopt abstinence or contraception measures during the study
3. Intake of an investigational drug within 1 month before the screening visit
4. Use of expectorants or drugs with expectorant effect within 2 days before randomization visit
5. Diagnosis of active tuberculosis, lung cancer, pulmonary fibrosis, acute pulmonary thromboembolism or any other respiratory condition that might, in the opinion of the investigator, compromise the safety of the patient or affect the interpretation of the results
6. Medical history of and/or illness (including laboratory abnormality) and/or treatment that in the investigator's opinion may interfere with the patient's safety, compliance, or study evaluations
7. Serum alanine aminotransferase and/or aspartate transaminase more than 3 times above the upper limit of normal at screening visit
8. Serum creatinine more than 3 times above the upper limit of normal at screening visit
9. Addiction to alcohol or drugs
10. Mental illness, or other reasons for non-cooperation in the investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- China (32):
  - Wuxi Peoples' Hospital affiliated to Nanjing Medical University, Wuxi, No. 299, Qing Yang Rd., Wuxi City, Jiangsu
  - Inner Mongolia Baogang Hospital, Baotou
  - Beijing Hospital, Beijing
  - Beijing Tongren Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University Shougang Hospital, Beijing
  - Jilin Province People's Hospital, Changchun
  - The First Bethune Hospital of Jilin University, Changchun
  - Chengdu Fifth People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Deyang People's Hospital, Deyang
  - Inner Mongolia People's Hospital, Hohhot
  - Jinhua city central hospital/Jinhua hospital ,School of Medicine,Zhejiang UNIVERSITY, Jinhua
  - Nanchang University-The Second Affiliated Hospital, Nanchang
  - Nanjing First Hospital, Nanjing
  - Zhongda Hospital, Southeast University - Pulmonology, Nanjing
  - Jiangxi Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - Minhang District Central Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Suining Central Hospital, Suining
  - First Hospital of Shanxi Medical University, Taiyuan
  - The First Hospital of Shanxi Medical University, Taiyuan
  - Tongji Hospital, Tongji Medical College of Huazhong University Science and Technology, Wuhan
  - Wuxi Peoples' Hospital affiliated to Nanjing Medical University, Wuxi
  - Yangzhou First People's Hospital, Yangzhou
  - General Hospital of Ningxia Medical University, Yinchuan
  - Affiliated Hospital of Guangdong Medical University - Respiration, Zhanjiang
  - The First People's Hospital of Zigong, Zigong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 21-June-2019 and 5-February-2021 in 28 sites in China.
Pre-assignment Details: Participants who met the inclusion and none of the exclusion criteria were enrolled to the study. All procedures were performed as per the trial flow chart.
Groups:
- N-Acetylcysteine: Participants received N-Acetylcysteine (NAC) 600 mg slow intravenous (IV) infusion twice daily (BD - morning and evening) for the 1-week treatment period.
- Ambroxol Hydrochloride: Participants received Ambroxol hydrochloride 30 mg slow intravenous infusion twice daily (morning and evening) for the 1-week treatment period.
- Placebo: Participants received placebo slow intravenous infusion twice daily (morning and evening) for the 1-week treatment period.
Period: Overall Study
Arm/Group | N-Acetylcysteine | Ambroxol Hydrochloride | Placebo
Started | 111 | 111 | 111
Modified ITT | 108 | 110 | 110
Completed | 96 | 95 | 97
Not Completed | 15 | 16 | 14
Not completed — Adverse Event | 4 | 2 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Lack of adherence to study medication | 0 | 0 | 1
Not completed — Physician Decision | 1 | 2 | 2
Not completed — Study subject withdrawal by parent or guardian | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 9 | 7
Not completed — Administration of rescue mucolytic | 0 | 0 | 1
Not completed — Reporting drug over temperature, patients plan to transfer to hospital, and discharge from hospital. | 2 | 3 | 0

BASELINE CHARACTERISTICS:
Population: mITT population - The Modified ITT (mITT) Population comprised all participants in the ITT population who received at least 1 dose or partial dose of the Investigational Medicinal Product (IMP).
Groups:
- N-Acetylcysteine: Participants received N-Acetylcysteine (NAC) 600 mg intravenous (IV) infusion twice daily (BD - morning and evening) for the 1-week treatment period.
- Ambroxol Hydrochloride: Participants received Ambroxol hydrochloride 30 mg intravenous infusion twice daily (morning and evening) for the 1-week treatment period.
- Placebo: Participants received placebo intravenous infusion twice daily (morning and evening) for the 1-week treatment period.
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Ambroxol Hydrochloride | Placebo | Total
Number analyzed (Participants) | 108 | 110 | 110 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.65) | 64.7 (12.76) | 64.5 (12.79) | 64.6 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 31 | 32 | 99
  Male | 72 | 79 | 78 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 108 | 110 | 110 | 328
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 7 of Mean Sputum Viscosity Score of NAC and Placebo
Description: The superiority of slow intravenous infusion of NAC to placebo in terms of change from baseline in sputum viscosity score was demonstrated. Sputum viscosity was assessed by ordinal categorical 4-point scales [0 = Liquid (normal viscosity), 1= Fluid (mildly increased viscosity), 2 = Viscous (moderately increased viscosity), 3 = Sticky (severely increased viscosity)] with 0 = best and 3= worst.
Time Frame: From baseline upto Day 7
Population: mITT population - The Modified ITT (mITT) Population comprised all participants in the ITT population who received at least 1 dose or partial dose of the IMP.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 108 | 110
Score | -1.2 (0.74) | -1.0 (0.78)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; For the superiority comparisons of NAC vs. placebo, the Bonferroni correction was used; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.24, Standard Deviation 0.763

2. Primary Outcome: Change From Baseline to Day 7 Treatment of Mean Expectoration Difficulty Score of NAC and Placebo
Description: The superiority of slow intravenous infusion of NAC 600 mg twice daily to placebo in terms of change from baseline in expectoration difficulty score was demonstrated. Expectoration difficulty was assessed by ordinal categorical 4-point scales [0 = No difficulty, 1 = Mild difficulty, 2 = Moderate difficulty, 3 = Marked difficulty] with 0 = best and 3 = worst.
Time Frame: From Baseline upto Day 7
Population: mITT population - The mITT population comprised all participants in the ITT population who received at least 1 dose or partial dose of the IMP.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 108 | 110
Score | -1.4 (0.78) | -1.1 (0.78)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; For the superiority comparisons of NAC vs. placebo, the Bonferroni correction was used; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.29, Standard Deviation 0.783

3. Secondary Outcome: Change From Baseline to Day 3 in Mean Sputum Viscosity Score of NAC and Placebo
Description: as for outcome 1
Time Frame: From Baseline to Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 108 | 110
Score | -0.6 (0.59) | -0.6 (0.64)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.239, Stratified Mann-Whitney U Statistic

4. Secondary Outcome: Change From Baseline to Day 3 in Mean Expectoration Difficulty Score of NAC and Placebo
Description: The superiority of slow intravenous infusion of NAC to placebo in terms of change from baseline in expectoration difficulty score was demonstrated. Expectoration difficulty was assessed by ordinal categorical 4-point scales [0 = No difficulty, 1 = Mild difficulty, 2 = Moderate difficulty, 3 = Marked difficulty] with 0 = best and 3 = worst.
Time Frame: From Baseline to Day 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 108 | 110
Score | -0.8 (0.61) | -0.7 (0.64)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; For the superiority comparisons of NAC vs. placebo, the Bonferroni correction was used; Test type: Superiority; p = 0.037, Stratified Mann-Whitney U Statistic

5. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 in Mean Sputum Color Score of NAC and Placebo
Description: The superiority of the slow intravenous infusion of NAC to placebo in terms of change from baseline in sputum color score was demonstrated. Sputum color was assessed by means of ordinal categorical 4-point scales [0 = Mostly white, 1= Mostly pale yellow, 2 = Mostly dark yellow, 3 = Very dark yellow /green] with 0 = best and 3= worst.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 108 | 110
Score
  Change from baseline to Day 3 | -0.5 (0.72) | -0.5 (0.82)
  Change from baseline to Day 7 | -0.8 (0.89) | -0.8 (0.97)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.093, Stratified Mann Whitney U Statistic
Statistical Analysis 2: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.118, Stratified Mann Whitney U Statistic

6. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 in Mean Cough Severity Score of NAC and Placebo
Description: The superiority of the slow intravenous infusion of NAC to placebo in terms of change from baseline in cough score was demonstrated. Cough score was assessed by means of ordinal categorical 4-point scales [0 = No cough, 1= Sporadic and mild cough, 2 = Moderate cough, 3 = Severe Cough] with 0 = best and 3= worst.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 108 | 110
Score
  Change from baseline to Day 3 | -0.4 (0.55) | -0.5 (0.60)
  Change from baseline to Day 7 | -0.8 (0.77) | -0.6 (0.72)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.022, Stratified Mann Whitney U Statistic
Statistical Analysis 2: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.110, Stratified Mann Whitney U Statistic

7. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 of Mean Sputum Volume of NAC and Placebo
Description: The superiority of the slow intravenous infusion of NAC to placebo in terms of change from baseline in sputum volume was demonstrated. Patients collected 24-hour sputum (morning to same time of the following morning) in a graduated cup and volume was expressed as mL/24h.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/24h
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 108 | 110
mL/24h
  Change from baseline to Day 3 | -1.601 (16.2611) | -4.144 (12.2348)
  Change from baseline to Day 7 | -9.405 (35.2191) | -7.391 (15.9992)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.022, Stratified Mann Whitney U Statistic
Statistical Analysis 2: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.402, Stratified Mann Whitney U Statistic

8. Secondary Outcome: Change From Baseline to Day 7 in Mean Sputum Viscosity Score of NAC and Ambroxol Hydrochloride
Description: The non-inferiority of NAC versus ambroxol in terms of change from baseline to Day 7 of mean sputum viscosity score was demonstrated. Sputum viscosity was assessed by ordinal categorical 4-point scales [0 = Liquid (normal viscosity), 1= Fluid (mildly increased viscosity), 2 = Viscous (moderately increased viscosity), 3 = Sticky (severely increased viscosity)] with 0 = best and 3= worst.
Time Frame: From baseline upto Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Ambroxol Hydrochloride
Number analyzed (Participants) | 108 | 110
Score | -1.2 (0.74) | -1.2 (0.78)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Ambroxol Hydrochloride; Test type: Non-Inferiority — Non-inferiority was declared if the one-sided confidence interval was within the interval; p = 0.002, Modified Mann-Whitney U Statistic; Probability scale treatment difference = 0.50, 97.5% CI 2-sided [0.43 to 1.00] — The point estimates of treatment differences in probability scale together with associated one-side confidence interval (97.5% or 98.75%) were computed according to Hochberg if both superiority contrasts were found statistically significant

9. Secondary Outcome: Change From Baseline to Day 7 in Mean Expectoration Difficulty Score of NAC and Ambroxol Hydrochloride
Description: The non-inferiority of NAC versus ambroxol in terms of change from baseline to Day 7 of mean expectoration difficulty score was demonstrated. Expectoration difficulty was assessed by ordinal categorical 4-point scales [0 = No difficulty, 1 = Mild difficulty, 2 = Moderate difficulty, 3 = Marked difficulty] with 0 = best and 3= worst
Time Frame: From Baseline upto Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | N-Acetylcysteine | Ambroxol Hydrochloride
Number analyzed (Participants) | 108 | 110
Score | -1.4 (0.78) | -1.3 (0.75)
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Ambroxol Hydrochloride; Test type: Non-Inferiority — Non-inferiority was declared if the one-sided confidence interval was within the interval; p < 0.001, Modified Mann-Whitney U Statistic; Probability scale treatment difference = 0.5, 98.75% CI 2-sided [0.45 to 1.00] — The point estimates of treatment differences in probability scale together with associated one-side confidence interval (97.5% or 98.75%) were computed according to Hochberg if both superiority contrasts were found statistically significant

10. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 in Mean Sputum Viscosity Score of Ambroxol Hydrochloride and Placebo
Description: The superiority of the slow intravenous infusion ambroxol hydrochloride to placebo in terms of change from baseline in sputum viscosity score was demonstrated. Sputum viscosity was assessed by ordinal categorical 4-point scales [0 = Liquid (normal viscosity), 1= Fluid (mildly increased viscosity), 2 = Viscous (moderately increased viscosity), 3 = Sticky (severely increased viscosity)] with 0 = best and 3= worst.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Ambroxol Hydrochloride | Placebo
Number analyzed (Participants) | 110 | 110
Score
  Change from baseline to Day 3 | -0.6 (0.55) | -0.6 (0.64)
  Change from baseline to Day 7 | -1.2 (0.78) | -1.0 (0.78)
Statistical Analysis 1: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.356, Modified Mann-Whitney U Statistic
Statistical Analysis 2: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.007, Modified Mann-Whitney U Statistic

11. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 in Mean Expectoration Difficulty Score of Ambroxol Hydrochloride and Placebo
Description: The superiority of the slow intravenous infusion of ambroxol hydrochloride to placebo in terms of change from baseline in expectoration difficulty score was demonstrated. Expectoration difficulty was assessed by ordinal categorical 4-point scales [0 = No difficulty, 1 = Mild difficulty, 2 = Moderate difficulty, 3 = Marked difficulty] with 0 = best and 3 = worst.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Ambroxol Hydrochloride | Placebo
Number analyzed (Participants) | 110 | 110
Score
  Change from baseline to Day 3 | -0.7 (0.57) | -0.7 (0.64)
  Change from baseline to Day 7 | -1.3 (0.75) | -1.1 (0.78)
Statistical Analysis 1: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.380, Modified Mann-Whitney U Statistic
Statistical Analysis 2: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.018, Modified Mann-Whitney U Statistic

12. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 in Mean Sputum Color Score of Ambroxol Hydrochloride and Placebo
Description: The superiority of slow intravenous infusion of ambroxol hydrochloride to placebo in terms of change from baseline in sputum color was demonstrated. Sputum color was assessed by means of ordinal categorical 4-point scales [0 = Mostly white, 1= Mostly pale yellow, 2 = Mostly dark yellow, 3 = Very dark yellow /green] with 0 = best and 3= worst.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Ambroxol Hydrochloride | Placebo
Number analyzed (Participants) | 110 | 110
Score
  Change from baseline to Day 3 | -0.5 (0.77) | -0.5 (0.82)
  Change from baseline to Day 7 | -0.9 (0.99) | -0.8 (0.97)
Statistical Analysis 1: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.366, Modified Mann-Whitney U Statistic
Statistical Analysis 2: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.027, Modified Mann-Whitney U Statistic

13. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 in Mean Cough Severity Score of Ambroxol Hydrochloride and Placebo
Description: The superiority of slow intravenous infusion of ambroxol hydrochloride to placebo in terms of change from baseline in cough score was demonstrated. Cough score was assessed by means of ordinal categorical 4-point scales [0 = No cough, 1= Sporadic and mild cough, 2 = Moderate cough, 3 = Severe Cough] with 0 = best and 3= worst.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Ambroxol Hydrochloride | Placebo
Number analyzed (Participants) | 110 | 110
Score
  Change from baseline to Day 3 | -0.4 (0.52) | -0.5 (0.60)
  Change from baseline to Day 7 | -0.7 (0.68) | -0.6 (0.72)
Statistical Analysis 1: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.052, Modified Mann-Whitney U Statistic
Statistical Analysis 2: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.058, Modified Mann-Whitney U Statistic

14. Secondary Outcome: Change From Baseline to Day 3 and to Day 7 in Mean Sputum Volume of Ambroxol Hydrochloride and Placebo
Description: The superiority of slow intravenous infusion of ambroxol hydrochloride to placebo in terms of change from baseline in mean sputum volume was demonstrated. Patients collected 24-hour sputum (morning to same time of the following morning) in a graduated cup and volume was expressed as mL/24h.
Time Frame: From Baseline upto Day 3 and Day 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/24h
Arm/Group | Ambroxol Hydrochloride | Placebo
Number analyzed (Participants) | 110 | 110
mL/24h
  Change from baseline to Day 3 | -4.53 (12.018) | -4.14 (12.235)
  Change from baseline to Day 7 | -9.73 (15.149) | -7.39 (15.999)
Statistical Analysis 1: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.309, Modified Mann-Whitney U Statistic
Statistical Analysis 2: Comparison: Ambroxol Hydrochloride vs Placebo; Test type: Superiority; p = 0.006, Modified Mann-Whitney U Statistic

15. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability of intravenous NAC 600 mg twice daily was demonstrated.
Time Frame: From screening to follow-up after the last administration of the investigational medicinal product (IMP) [assessed up to 19 months]
Population: The safety population included all subjects who provided informed consent and received at least 1 dose or partial dose of the IMP. Subjects were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | N-Acetylcysteine | Ambroxol Hydrochloride | Placebo
Number analyzed (Participants) | 108 | 110 | 110
Participants
  At least one AE | 82 | 76 | 71
  At least one TEAE | 67 | 66 | 58
  At least one IMP-related TEAE | 11 | 11 | 0
  At least one TEAE leading to drug withdrawal | 5 | 2 | 3
  At least one TEAE leading to drug interruption | 0 | 0 | 1
  At least one TEAE leading to fatal outcome | 1 | 0 | 0
  At least one severe TEAE | 5 | 4 | 7
  At least one TEAE of COVID-19 | 0 | 0 | 0
  At least one SAE | 2 | 5 | 7
  At least one TESAE | 2 | 5 | 7
  At least one TESAE leading to drug withdrawal | 1 | 1 | 1
  At least one TESAE leading to drug interruption | 0 | 0 | 1
  At least one TESAE leading to fatal outcome | 1 | 0 | 0
  At least one TESAE of COVID-19 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening to follow-up after the last administration of the investigational medicinal product (IMP) [assessed up to 19 months].
Description: The Safety Population has been considered to report AEs. It comprised 328 subjects who provided informed consent and received at least 1 dose or partial dose of the IMP.
Arm/Group | N-Acetylcysteine | Ambroxol Hydrochloride | Placebo
All-Cause Mortality (participants affected / at risk) | 1/108 | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 2/108 | 5/110 | 7/110
Other Adverse Events (participants affected / at risk) | 67/108 | 66/110 | 58/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-Acetylcysteine (N=108) | Ambroxol Hydrochloride (N=110) | Placebo (N=110)
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Non-small lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Congenital cerebrovascular anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=108) | Ambroxol Hydrochloride (N=110) | Placebo (N=110)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Chronic gastritis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroptosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoplakia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (13) | 9 (9) | 9 (9)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Asymptomatic bacteriuria (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Urinary occult blood positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Beta 2 microglobulin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Carbohydrate antigen 19-9 increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Carbon dioxide increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Carcinoembryonic antigen increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram Q wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid factor increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Tumour marker increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 2 (2) | 3 (3) | 4 (4)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 2 (2) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 2 (2) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gallbladder cholesterolosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic calcification (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (3) | 2 (2) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cor pulmonale chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 3 (3) | 3 (3)
Renal cyst (Renal and urinary disorders) | 1 (1) | 6 (6) | 3 (3)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal meningeal cyst (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 1 (1) | 2 (2)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial stiffness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 3 (4)
Calculus prostatic (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 3 (3) | 2 (2)
Goitre (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Secondary hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal leukoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Immunodeficiency (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains confidential information of Zambon S.p.A. Do not copy or distribute without written permission from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03843541/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03843541/SAP_001.pdf